CLINICAL TRIAL: NCT00714844
Title: Waist Circumference Reduction After Insulin Detemir Treatment in Type 2 Diabetes Patients Previously Treated With NPH Insulin
Brief Title: Insulin Detemir and Waist Circumference
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Susanna Morano, University of Roma La Sapienza, Policlinico Umberto I, Dpt Scienze Cliniche
Other Study IDs: PolUmbI-DptSClin-Det1
Record Dates: First submitted 2008-07-07; First posted 2008-07-14 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-04

CONDITIONS: Type 2 Diabetes
Keywords: insulin therapy; insulin detemir; waist circumference
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to investigate the weight-sparing effect of detemir and assess glycemic control and treatment satisfaction when switching from NPH to detemir, to improve metabolic control.

ELIGIBILITY:
Inclusion Criteria:

* Duration of type 2 diabetes for at least 12 months
* BMI <40 kg/m2
* HbA1c >7.5%
* Requiring basal insulin replacement and previously treated with NPH insulin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetic patients accessing the Diabetologic Centre
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

REFERENCES:
- [Derived] Mandosi E, Fallarino M, Rossetti M, Gatti A, Morano S. Waist circumference reduction after insulin detemir therapy in type 2 diabetes patients previously treated with NPH. Diabetes Res Clin Pract. 2009 May;84(2):e18-20. doi: 10.1016/j.diabres.2009.02.006. Epub 2009 Mar 17. PMID 19297054